CLINICAL TRIAL: NCT05730829
Title: Pain Informed Movement for People With Knee Osteoarthritis: A Pilot and Feasibility Randomized Controlled Trial
Brief Title: Pain Informed Movement for People With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Boston University (Other); University of Melbourne (Other); University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HiREB 15700
Record Dates: First submitted 2023-02-06; First posted 2023-02-16 (Actual); Results first posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2024-11

CONDITIONS: Knee Osteoarthritis
Keywords: pain modulation; mind-body exercise
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Educational Status

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pain Informed Movement and pain neuroscience education (Experimental): Participants will receive a twice weekly, 8 week in-person group exercise program, consisting of exercise instruction (75 minutes) and pain neuroscience education (PNE) videos (20 to 30 minutes/week for the first 4 weeks). During the exercise sessions, the educational components and concepts such as mindfulness, muscle tension regulation, and breathing techniques will be applied by the instructor. A third home session (weekly) will be facilitated by exercise handout sheets. The exercise component will be delivered by an experienced yoga teacher that has been extensively trained. The PNE video component will cover the following topics: The purpose of pain, neurophysiological changes of pain, movement guidelines when pain persists, and self-care techniques to impact neurophysiology and support moving with ease that include breath awareness and regulation, muscle tension regulation, awareness of pain related thoughts and emotions, relaxation, and body awareness.
  Interventions: Other: pain informed movement; Other: Pain Neuroscience Education (PNE)
- Standard neuromuscular exercise and OA education (Active Comparator): Participants in this group will receive an 8-week in-person group exercise program held twice weekly, in which they will receive exercise instructions (60 minutes) and standard osteoarthritis (OA) education (15 to 20 minutes/week for the first 4 weeks). A third home session (weekly) will be facilitated by exercise handout sheets. The exercise component (i.e., the specific movements) of this group will be similar to those of the other group without the added techniques of breath awareness and regulation, muscle tension regulation, awareness of pain related thoughts and emotions, relaxation, and body awareness. The standard OA education videos will cover the following topics: common OA symptoms, risk factors associated with knee OA, and the effects of exercise and self-management tips. The exercise and education components will be delivered by a physiotherapist in the research team.
  Interventions: Other: standard neuromuscular exercise; Other: Standard osteoarthritis (OA) education

INTERVENTIONS:
Other: pain informed movement — group classes twice weekly for 8 weeks of neuromuscular exercise in combination with mind-body techniques such as breath regulation, muscle tension regulation, relaxation, mindfulness, awareness of pain related thoughts and emotions.
  Arms: Pain Informed Movement and pain neuroscience education
Other: standard neuromuscular exercise — group classes twice weekly for 8 weeks of neuromuscular exercise.
  Arms: Standard neuromuscular exercise and OA education
Other: Pain Neuroscience Education (PNE) — The pain neuroscience education (PNE) will be delivered in videos addressing concepts such as the purpose of pain, neurophysiological changes of pain, movement guidelines when pain persists, and self-care techniques to impact neurophysiology and support moving with ease that include breath awareness and regulation, muscle tension regulation, awareness of pain related thoughts and emotions, relaxation, and body awareness.
  Arms: Pain Informed Movement and pain neuroscience education
Other: Standard osteoarthritis (OA) education — The standard osteoarthritis (OA) education will address the following topics, OA prevalence, risk factors, symptoms, diagnosis, treatment, role of exercise, surgery, self-management
  Arms: Standard neuromuscular exercise and OA education

SUMMARY:
The goal of this clinical trial is to compare a pain informed movement program to standard neuromuscular exercise in people with knee osteoarthritis. The main question it aims to answer are:

1. Are the two interventions a) pain informed movement program plus pain neuroscience education and b) neuromuscular exercise plus standard osteoarthritis education feasible in terms of recruitment, treatment adherence, timelines, data collection procedures, patient follow-up, and resources required?
2. Is there a difference in patient's satisfaction and acceptability of the two programs?
3. Are there any differences in the potential effects of the two programs on subjective pain measures, self-reported function, quality of life, functional leg strength, nervous system pain modulation, brain derived neurotrophic factor and nerve growth factor levels, and psychological factors?

DETAILED DESCRIPTION:
It is critical to understand the underlying mechanism of knee osteoarthritis (OA) pain in order to effectively manage knee OA. It has become clear that alterations in central and peripheral nervous system functioning occurs in people with knee OA and pain sensitization is a common feature. Descending modulation from the central nervous system can facilitate or inhibit nociception. Endogenous pain modulation through the descending system is an important factor as its dysregulation has significant ramifications in pain facilitation and promotion of chronic pain development and maintenance at all levels of the nervous system. The current guidelines lack focus on how to effectively manage it, which is a potential reason for why the current methods in conservative management of knee OA pain are only moderately effective. Mind-body approaches are uniquely positioned to potentially reverse the sensitization, induce positive neuroplastic changes, and improve descending pain modulation resulting in decreased pain intensity in many chronic pain populations. This study involves an exercise program which the investigators call 'Pain Informed Movement' that includes evidence-based exercises combined with mind-body techniques and pain neuroscience education. The data from this phase will be used to inform a multi-site randomized controlled trial (RCT) to assess the program's effectiveness with the primary outcome of change in pain severity mediated by change in descending pain modulation.

Exercise is regularly used as a first-line management option for knee OA, and its use is supported by high quality evidence to improve pain and function. Clinical practice guidelines for people with knee OA recommend the use of aerobic and strength training for the reduction of pain and improved physical function. Currently, one of the key components of conservative management of knee OA often implemented by clinicians is a type of exercise called neuromuscular exercise, which aims at improving sensorimotor control and the functionality of the knee joint by addressing movement in all three movement planes. Previous research has showed that the neuromuscular exercise programs designed specifically for knee OA can reduce pain, improve function, alter knee biomechanics, and improve the muscle-activation patterns of the surrounding knee musculature. While exercise is the first line treatment for knee OA and can lead to improvements in physical function and pain, it is important to highlight that it has a moderate effect, which may be short term.

In recent years multiple guidelines for non-surgical management of knee OA have begun to include mind-body therapies, such as yoga or tai-chi, as conditional or core treatment recommendations. Mind-body therapies can lead to pain reductions and improvement of function through various techniques. For instance, breathing exercises including breath awareness and regulation can activate the parasympathetic nervous system and decrease the danger signals of pain, leading to improvement of pain levels. Meditative breathing can lead to reductions in pain levels by modulating the somatosensory cortex. Relaxation techniques focused on relaxing the muscles that become tense as a result of pain and by association can re-enforce or aggravate pain, can influence the pain experience by reversing that association. Mindfulness meditation and mindful movement which can lead to a switch from sensory pain to the interoceptive awareness of the movements of the different body parts, resulting in reduced muscle tension, improvements in postural stability and proprioception, and reductions in pain levels. Mind-body therapies also lead to improvement of psychological factors such as depression, anxiety, pain catastrophizing, increasing pain acceptance, changing patients' relationships to their pain, which in turn lead to reductions in pain levels. The positive effects of mindfulness practices have been reported to last in longer-term follow ups such as 15 months, and 3 years.

Education is another core component recommended by clinical guidelines and known to be effective particularly when combined with exercise. Pain Neuroscience education (PNE) is an alternative technique of teaching patients about pain and how to rethink and re-evaluate the way pain is viewed. The use of PNE in physical therapy interventions has been steadily increasing due to its positive effects on pain and function in many chronic pain patient populations. PNE includes an explanation of the neurophysiology of pain and its process by the nervous system. This includes how pain can be modulated through upregulation or downregulation of signals to increase or decrease the pain experience and that these changes are not necessarily related to tissue damage, particularly when pain becomes chronic. PNE also provides information regarding the influence of various psychosocial aspects. By offering avenues to reconceptualize pain as a threat to the body and movement as imminent danger, patients may become more willing to participate in physical activity and tolerate slight increases in pain and discomfort.

In contrast standard OA education is the traditional and most widely used educational model in people with knee OA, focuses heavily on a pathoanatomical perspective of pain referring mainly to anatomy, biomechanics, and patho-anatomy of OA and the knee joint.

Given the importance of finding effective management strategies for pain modulation in people with knee OA, there is a need to further our understanding of the impact of evidence-based exercise combined with mind-body techniques (e.g., breathing exercises and mindfulness) with PNE on pain mechanisms.

The study is a pilot RCT with a nested qualitative component. The study will be guided by the Conceptual Framework for Defining Feasibility and Pilot studies and the Standard Protocol Items: Recommendations for Intervention Trials.

Study Population

A sample of 66 adults will be sought. The sample size is based on the primary outcome of complete follow-up using the confidence interval method for calculating sample size in pilot trials. 90% follow-up rate is the aim but the trial will be considered successful if 81% is achieved. To achieve a margin of error of 9%, with 10% added for attrition, 66 participants is required.

Recruitment Participants will be recruited through the email lists of the McMaster Physical Activity Centre of Excellence (PACE) community and the McMaster Institute for Research on Aging (MIRA) newsletter. Postings will be placed on both PACE and MIRA social media pages. In addition, the study poster will be placed on other social media channels (i.e., Twitter, Facebook advertisements). In addition, flyers will be placed in local orthopaedic surgeon, Rheumatologist and Physiatrists offices. Physicians will provide potential participants with a one-page study information sheet in lay language. If interested, potential participants can then contact the research team through the contact information provided in the flyer.

Setting The in-person 8-week exercise program will be held twice weekly at McMaster University's Physical Activity Centre of Excellence (PACE) located in the Ivor-Wynne Centre or in one of two local community churches. Participants will complete the pain assessment, and have blood drawn at PACE by PACE staff who are certified phlebotomists.

Assessment As part of participation in the study, participants will be asked to attend an assessment at the beginning of the study, and once again upon completing the 8-week exercise program. Participants will conditioned undergo pain modulation (CPM) and mechanical temporal summation testing, and the 30 Second Sit to Stand Test to determine leg strength and endurance. Lastly, participants will have their blood drawn (fasting) at the beginning and end of the study. Participants will then be asked to complete a series of questionnaires about their pain and mood.

Interventions Twice weekly group exercise sessions will be 75 minutes for the intervention group and 60 minutes in duration for the control group. The intervention arm class is slightly longer due to the detailed delivery of instructions for the techniques during the class. Participants will be given instructions to complete these exercises at home at least one other time during the week for the same duration. Participants will receive education videos that are ~15-20 minutes each week, for up to 4 weeks.

Pain Informed Movement and PNE - During the neuromuscular exercise sessions, the PNE components and concepts such as mindfulness, muscle tension regulation, and breathing techniques will be applied by the instructor.

Neuromuscular exercise and standard OA education - The exercise component (i.e., the specific movements) of this group will be similar to those of the intervention group without the added mind-body techniques.

Randomization and allocation concealment Participants will be randomized with an allocation ratio of 1:1 into one of two treatment groups (Pain informed movement and PNE versus neuromuscular exercise and standard OA education) using a REDCap randomization module. Following consent and completion of baseline assessment, the assessor (different person than the recruiter) will log in to the website, open the participants' identification record and click on the randomize button. Randomization will be blocked and this process will ensure allocation concealment. As allocation concealment occurs following the baseline assessment, the assessors will be blinded at baseline and follow up assessment. Blinding of instructors is generally not possible in studies of physical interventions (i.e., exercise). Participants will be blinded to study hypotheses and the two treatment groups. As both arms of the study are providing exercise based interventions and education, participants will be provided limited details of each intervention arm so as to blind them from knowing which is the intervention and which is the control. This will help minimize any bias that occurs by knowledge of group assignment and perception of treatment effects.

Exit Survey and Focus Group In addition to the primary and secondary outcomes, a satisfaction survey will be conducted at the end of the program to evaluate the a priori feasibility criteria. Participants who indicated upon initially consenting to the study that would like to participate in a focus group, will be contacted. Qualitative data collection will be used to explore participants experience and perceptions of the feasibility and acceptability of the program. A focus group will be conducted using audio or video recording (using Zoom), lasting between 45-60 minutes.

ELIGIBILITY:
Inclusion Criteria:

* - ≥40 years of age with diagnosis of knee osteoarthritis (OA) by a physician OR;
* ≥45 years of age and having activity-related knee joint pain with or without morning stiffness lasting 30 minutes (NICE criteria)
* Having an average pain intensity of 3/10 on a numeric pain scale on most days of the past month

Exclusion Criteria:

* Cannot communicate in English;
* Has inflammatory arthritis or other systemic conditions;
* Have had lower limb trauma or surgery within the past 6 months;
* Have participated in a knee OA exercise program in the prior 3 months;
* Have had any injection in the index knee within 3-months prior to baseline assessment
* Does not have regular access to the internet
* Inability to get up and down from the floor independently
* Use of mobility aids
* Currently participating in any other drug/device/exercise clinical trial related to OA
* Planned absences (e.g., trips away) of >1 week
* Currently receiving other forms of care for knee OA pain (e.g., from a physiotherapist, chiropractor, athletic therapist, kinesiologist)
* Does not meet screening for safe participation in exercise according to the Get Active questionnaire from the Canadian Society for Exercise Physiology

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2023-04-03 (Actual); Primary Completion 2024-12-03 (Actual); Study Completion 2024-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Carlesso, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fingleton C, Smart K, Moloney N, Fullen BM, Doody C. Pain sensitization in people with knee osteoarthritis: a systematic review and meta-analysis. Osteoarthritis Cartilage. 2015 Jul;23(7):1043-56. doi: 10.1016/j.joca.2015.02.163. Epub 2015 Mar 5. PMID 25749012
- [Background] Carlesso LC, Segal NA, Frey-Law L, Zhang Y, Na L, Nevitt M, Lewis CE, Neogi T. Pain Susceptibility Phenotypes in Those Free of Knee Pain With or at Risk of Knee Osteoarthritis: The Multicenter Osteoarthritis Study. Arthritis Rheumatol. 2019 Apr;71(4):542-549. doi: 10.1002/art.40752. Epub 2019 Feb 7. PMID 30307131
- [Background] Neogi T, Frey-Law L, Scholz J, Niu J, Arendt-Nielsen L, Woolf C, Nevitt M, Bradley L, Felson DT; Multicenter Osteoarthritis (MOST) Study. Sensitivity and sensitisation in relation to pain severity in knee osteoarthritis: trait or state? Ann Rheum Dis. 2015 Apr;74(4):682-8. doi: 10.1136/annrheumdis-2013-204191. Epub 2013 Dec 18. PMID 24351516
- [Background] Petersen KK, Graven-Nielsen T, Simonsen O, Laursen MB, Arendt-Nielsen L. Preoperative pain mechanisms assessed by cuff algometry are associated with chronic postoperative pain relief after total knee replacement. Pain. 2016 Jul;157(7):1400-1406. doi: 10.1097/j.pain.0000000000000531. PMID 27331347
- [Background] Fransen M, McConnell S, Harmer AR, Van der Esch M, Simic M, Bennell KL. Exercise for osteoarthritis of the knee: a Cochrane systematic review. Br J Sports Med. 2015 Dec;49(24):1554-7. doi: 10.1136/bjsports-2015-095424. Epub 2015 Sep 24. PMID 26405113
- [Background] Anwer S, Alghadir A, Brismee JM. Effect of Home Exercise Program in Patients With Knee Osteoarthritis: A Systematic Review and Meta-analysis. J Geriatr Phys Ther. 2016 Jan-Mar;39(1):38-48. doi: 10.1519/JPT.0000000000000045. PMID 25695471
- [Background] Rice D, McNair P, Huysmans E, Letzen J, Finan P. Best Evidence Rehabilitation for Chronic Pain Part 5: Osteoarthritis. J Clin Med. 2019 Oct 24;8(11):1769. doi: 10.3390/jcm8111769. PMID 31652929
- [Background] Yarnitsky D. Role of endogenous pain modulation in chronic pain mechanisms and treatment. Pain. 2015 Apr;156 Suppl 1:S24-S31. doi: 10.1097/01.j.pain.0000460343.46847.58. PMID 25789433
- [Background] Damien J, Colloca L, Bellei-Rodriguez CE, Marchand S. Pain Modulation: From Conditioned Pain Modulation to Placebo and Nocebo Effects in Experimental and Clinical Pain. Int Rev Neurobiol. 2018;139:255-296. doi: 10.1016/bs.irn.2018.07.024. Epub 2018 Aug 14. PMID 30146050
- [Background] Hassed C. Mind-body therapies--use in chronic pain management. Aust Fam Physician. 2013 Mar;42(3):112-7. PMID 23529519
- [Background] Kolasinski SL, Neogi T, Hochberg MC, Oatis C, Guyatt G, Block J, Callahan L, Copenhaver C, Dodge C, Felson D, Gellar K, Harvey WF, Hawker G, Herzig E, Kwoh CK, Nelson AE, Samuels J, Scanzello C, White D, Wise B, Altman RD, DiRenzo D, Fontanarosa J, Giradi G, Ishimori M, Misra D, Shah AA, Shmagel AK, Thoma LM, Turgunbaev M, Turner AS, Reston J. 2019 American College of Rheumatology/Arthritis Foundation Guideline for the Management of Osteoarthritis of the Hand, Hip, and Knee. Arthritis Care Res (Hoboken). 2020 Feb;72(2):149-162. doi: 10.1002/acr.24131. Epub 2020 Jan 6. PMID 31908149
- [Background] Bannuru RR, Osani MC, Vaysbrot EE, Arden NK, Bennell K, Bierma-Zeinstra SMA, Kraus VB, Lohmander LS, Abbott JH, Bhandari M, Blanco FJ, Espinosa R, Haugen IK, Lin J, Mandl LA, Moilanen E, Nakamura N, Snyder-Mackler L, Trojian T, Underwood M, McAlindon TE. OARSI guidelines for the non-surgical management of knee, hip, and polyarticular osteoarthritis. Osteoarthritis Cartilage. 2019 Nov;27(11):1578-1589. doi: 10.1016/j.joca.2019.06.011. Epub 2019 Jul 3. PMID 31278997
- [Background] Pearson N, Prosko S, Sullivan M, Taylor MJ. White Paper: Yoga Therapy and Pain-How Yoga Therapy Serves in Comprehensive Integrative Pain Management, and How It Can Do More. Int J Yoga Therap. 2020 Jan 1;30(1):117-133. doi: 10.17761/2020-D-19-00074. PMID 32412808
- [Background] Busch V, Magerl W, Kern U, Haas J, Hajak G, Eichhammer P. The effect of deep and slow breathing on pain perception, autonomic activity, and mood processing--an experimental study. Pain Med. 2012 Feb;13(2):215-28. doi: 10.1111/j.1526-4637.2011.01243.x. Epub 2011 Sep 21. PMID 21939499
- [Background] Ma X, Yue ZQ, Gong ZQ, Zhang H, Duan NY, Shi YT, Wei GX, Li YF. The Effect of Diaphragmatic Breathing on Attention, Negative Affect and Stress in Healthy Adults. Front Psychol. 2017 Jun 6;8:874. doi: 10.3389/fpsyg.2017.00874. eCollection 2017. PMID 28626434
- [Background] Russo MA, Santarelli DM, O'Rourke D. The physiological effects of slow breathing in the healthy human. Breathe (Sheff). 2017 Dec;13(4):298-309. doi: 10.1183/20734735.009817. PMID 29209423
- [Background] Schlereth T, Birklein F. The sympathetic nervous system and pain. Neuromolecular Med. 2008;10(3):141-7. doi: 10.1007/s12017-007-8018-6. Epub 2007 Nov 8. PMID 17990126
- [Background] Majeed MH, Ali AA, Sudak DM. Mindfulness-based interventions for chronic pain: Evidence and applications. Asian J Psychiatr. 2018 Feb;32:79-83. doi: 10.1016/j.ajp.2017.11.025. Epub 2017 Dec 5. PMID 29220782
- [Background] van Doormaal MCM, Meerhoff GA, Vliet Vlieland TPM, Peter WF. A clinical practice guideline for physical therapy in patients with hip or knee osteoarthritis. Musculoskeletal Care. 2020 Dec;18(4):575-595. doi: 10.1002/msc.1492. Epub 2020 Jul 9. PMID 32643252
- [Background] Louw A, Puentedura EJ, Reed J, Zimney K, Grimm D, Landers MR. A controlled clinical trial of preoperative pain neuroscience education for patients about to undergo total knee arthroplasty. Clin Rehabil. 2019 Nov;33(11):1722-1731. doi: 10.1177/0269215519857782. Epub 2019 Jun 19. PMID 31213078
- [Background] Louw A, Diener I, Butler DS, Puentedura EJ. The effect of neuroscience education on pain, disability, anxiety, and stress in chronic musculoskeletal pain. Arch Phys Med Rehabil. 2011 Dec;92(12):2041-56. doi: 10.1016/j.apmr.2011.07.198. PMID 22133255
- [Background] Wijma AJ, van Wilgen CP, Meeus M, Nijs J. Clinical biopsychosocial physiotherapy assessment of patients with chronic pain: The first step in pain neuroscience education. Physiother Theory Pract. 2016 Jul;32(5):368-84. doi: 10.1080/09593985.2016.1194651. Epub 2016 Jun 28. PMID 27351769
- [Background] Eldridge SM, Chan CL, Campbell MJ, Bond CM, Hopewell S, Thabane L, Lancaster GA; PAFS consensus group. CONSORT 2010 statement: extension to randomised pilot and feasibility trials. BMJ. 2016 Oct 24;355:i5239. doi: 10.1136/bmj.i5239. PMID 27777223
- [Background] Chan AW, Tetzlaff JM, Altman DG, Laupacis A, Gotzsche PC, Krleza-Jeric K, Hrobjartsson A, Mann H, Dickersin K, Berlin JA, Dore CJ, Parulekar WR, Summerskill WS, Groves T, Schulz KF, Sox HC, Rockhold FW, Rennie D, Moher D. SPIRIT 2013 statement: defining standard protocol items for clinical trials. Ann Intern Med. 2013 Feb 5;158(3):200-7. doi: 10.7326/0003-4819-158-3-201302050-00583. PMID 23295957
- [Background] Thabane L, Ma J, Chu R, Cheng J, Ismaila A, Rios LP, Robson R, Thabane M, Giangregorio L, Goldsmith CH. A tutorial on pilot studies: the what, why and how. BMC Med Res Methodol. 2010 Jan 6;10:1. doi: 10.1186/1471-2288-10-1. PMID 20053272

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: NA. we did not have any significant event prior to assignment of participants to an arm.
Groups:
- Pain Informed Movement and Pain Neuroscience Education: Participants will engage in a twice-weekly, 8-week in-person group exercise program, combining neuromuscular exercise and mind-body techniques. Each session includes 75 minutes of exercise instruction and, during the first four weeks, 20 to 30 minutes of Pain Neuroscience Education (PNE) videos. A third weekly home session will be supported by exercise handouts. The exercise component will be led by an experienced yoga instructor trained extensively in pain-informed movement, incorporating techniques such as breath regulation, muscle tension regulation, relaxation, mindfulness, and awareness of pain-related thoughts and emotions.
  The PNE videos will cover key topics: the purpose of pain, neurophysiological changes in pain, movement strategies when pain persists, and self-care techniques to influence neurophysiology. These include breath awareness, muscle tension regulation, and relaxation methods aimed at supporting movement with greater ease while fostering body awareness and emotional regulation.
Period: Overall Study
Arm/Group | Pain Informed Movement and Pain Neuroscience Education | Standard Neuromuscular Exercise and OA Education
Started | 34 | 35
Completed | 28 | 31
Not Completed | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pain Informed Movement and Pain Neuroscience Education | Standard Neuromuscular Exercise and OA Education | Total
Number analyzed (Participants) | 28 | 31 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (9) | 62 (10) | 63 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 19 | 42
  Male | 5 | 12 | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 25 | 28 | 53
  Asian | 2 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Follow up
Description: The follow-up rate is calculated as the number (percentage) of participants who completed the study out of those who completed the baseline assessment.
Time Frame: 8 weeks
Population: This is the number of participants at baseline who completed the baseline assessments and enrolled in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Pain Informed Movement and Pain Neuroscience Education | Standard Neuromuscular Exercise and OA Education
Number analyzed (Participants) | 34 | 35
Participants | 28 | 31

2. Secondary Outcome: Number of Participants Who Considered the Program Useful and Very Useful
Description: the number of participants who found the program useful or very useful. Participants rated the program's usefulness on a Likert scale, ranging from "Not useful at all" to "Very useful." The final count reflects those who selected either of the top two response categories, indicating a positive perception of the program's value.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pain Informed Movement and Pain Neuroscience Education | Standard Neuromuscular Exercise and OA Education
Number analyzed (Participants) | 28 | 31
Participants | 25 | 29

3. Secondary Outcome: Number of Participants Who Considered the Program Frequent Enough
Description: This outcome measure represents the number of participants who rated the program's frequency as "Frequent enough" on a 5-point Likert scale. The scale ranged from "Not frequent enough" to "Frequent enough," capturing participants' satisfaction with the program's scheduling.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pain Informed Movement and Pain Neuroscience Education | Standard Neuromuscular Exercise and OA Education
Number analyzed (Participants) | 28 | 31
Participants | 24 | 25

4. Secondary Outcome: Number of Participants Who Considered the Educational Session Frequency Enough
Description: This outcome measure represents the number of participants who rated the frequency of the educational sessions as "Frequent enough" on a 5-point Likert scale. The scale ranged from "Not frequent enough" to "Frequent enough," assessing participants' satisfaction with the scheduling of the sessions.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pain Informed Movement and Pain Neuroscience Education | Standard Neuromuscular Exercise and OA Education
Number analyzed (Participants) | 28 | 31
Participants | 24 | 25

5. Secondary Outcome: Rate of Recruitment Measured by Number of People Recruited in a Year
Description: recruitment rate is a minimum of 40 people in a year
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Pain Informed Movement and Pain Neuroscience Education | Standard Neuromuscular Exercise and OA Education
Number analyzed (Participants) | 34 | 35
Participants | 28 | 31

6. Secondary Outcome: Percentage of Participants Who Did Not Find the Study Procedures Burdensome (Questionnaires, Tests, Blood Draws) Measured on 0-10 Scale
Description: This outcome measure represents the percentage of participants who rated the program's burdensomeness as zero, using a scale from 0 ("No burden at all") to 10 ("Very much a burden"). Participants who provided a low burden rating (≤3/10) are included in this percentage, indicating that they did not perceive the program as burdensome.
Time Frame: 8 weeks
Population: The percentage of the participants per arm who did not find the study procedures burdensome.
Measure: Number; unit: percentage of the participants
Arm/Group | Pain Informed Movement and Pain Neuroscience Education | Standard Neuromuscular Exercise and OA Education
Number analyzed (Participants) | 28 | 31
percentage of the participants
  Burden of questionnaires | 69 | 87
  Burden of physical assessments | 83 | 94

7. Secondary Outcome: Rate of Adherence Measured by Number of Sessions Attended and Home Sessions Completed
Description: This outcome measure evaluates adherence to the program by calculating the number of sessions attended in-person and the number of home sessions completed by participants. The rate of adherence is determined by the proportion of sessions attended and completed relative to the total number of scheduled sessions.
Time Frame: 8 weeks
Population: This is the total number of possible sessions for each group (16 sessions * Number of participants per group)
Measure: Number; unit: number of sessions attended in each grou
Units Other Than Participants: Number of sessions
Arm/Group | Pain Informed Movement and Pain Neuroscience Education | Standard Neuromuscular Exercise and OA Education
Number analyzed (Participants) | 28 | 31
Number analyzed (Number of sessions) | 448 | 496
number of sessions attended in each grou | 396 | 425

8. Secondary Outcome: Rate of Adverse Events Measured by Question Regarding Symptom Flare and Seeking Treatment
Description: measured as any problem that lasts for >2 days and/or causes the participant to seek other treatment
Time Frame: 8 weeks
Measure: Number; unit: Number of adverse events
Arm/Group | Pain Informed Movement and Pain Neuroscience Education | Standard Neuromuscular Exercise and OA Education
Number analyzed (Participants) | 28 | 31
Number of adverse events | 0 | 0

9. Other Pre Specified Outcome: Modified Charlson Comorbidity Index
Description: to assesses the presence of comorbidities minimum score = 0, maximum = 20 with higher scores indicating greater severity.
Time Frame: baseline
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Participant Characteristics
Description: Ethnicity
Time Frame: baseline
Population: Ethnicity: Caucasian n (%)
Measure: Count of Participants; unit: Participants
Arm/Group | Pain Informed Movement and Pain Neuroscience Education | Standard Neuromuscular Exercise and OA Education
Number analyzed (Participants) | 28 | 31
Participants | 25 | 28

11. Other Pre Specified Outcome: Weight
Description: Weight
Time Frame: baseline and 8 weeks
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Number of Participants With Medication Use
Description: This outcome measure represents the number of participants who reported taking any medication on a regular schedule. Medication use was assessed with a yes/no response, where participants indicated whether they consistently take any prescribed or over-the-counter medications.
Time Frame: baseline and 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pain Informed Movement and Pain Neuroscience Education | Standard Neuromuscular Exercise and OA Education
Number analyzed (Participants) | 28 | 31
Participants
  Baseline | 18 | 9
  8 weeks | 16 | 10

13. Other Pre Specified Outcome: Perspectives on Knee Replacement Surgery
Description: Three questions will be asked: 1. Are your knee symptoms so severe that you wish to undergo knee replacement surgery? 2. Do you think knee replacement surgery is eventually inevitable? 3. In your opinion, what factor(s) can lead to better outcomes after knee replacement surgery?
Time Frame: baseline and 8 weeks
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Other Painful Body Parts
Description: Using a body diagram, participants will be asked to indicate any other areas where they experience pain
Time Frame: baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: mean number of painful joints
Arm/Group | Pain Informed Movement and Pain Neuroscience Education | Standard Neuromuscular Exercise and OA Education
Number analyzed (Participants) | 28 | 31
mean number of painful joints
  Baselin | 3.6 (2.8) | 2.9 (1.9)
  8 weeks | 4 (3.9) | 2.36 (1.5)

15. Other Pre Specified Outcome: Mechanical Temporal Summation (TS)
Description: A 512mN weighted probe was applied at the volar wrist opposite to the index knee. Participants were asked to rate their pain on a scale from 0 (no pain) to 100 (worst imaginable pain). Then, the same stimulus was applied 10 times at a rate of 1 per second (guided by a metronome), and participants were again asked to rate their pain. Temporal Summation (TS) was defined as present if the pain rating after the repeated stimuli was higher than the initial pain rating. The TS score was calculated as the difference between the pain rating after the repeated stimuli and the initial pain rating at each timepoint.
Time Frame: baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pain Informed Movement and Pain Neuroscience Education | Standard Neuromuscular Exercise and OA Education
Number analyzed (Participants) | 28 | 31
score on a scale
  Follow-up | 1.6 (1.4) | 1.7 (1.4)
  Baseline | 1.8 (1.6) | 2.02 (1.54)

16. Other Pre Specified Outcome: Conditioned Pain Modulation (CPM) Measured With PPT Test Stimulus and Conditioning Stimulus of Forearm Ischemia
Description: First stimulus of pressure pain threshold is delivered, next ischemic forearm test is conducted to a 4/10 and then PPT is repeated. An index will be created by calculating the percent efficiency of CPM (%CPM) as PPT2/PPT1, multiplied by 100; whereby %CPM ≤ 100 indicates inefficient pain modulation CPM. There are no standard minimum or maximum values.
Time Frame: baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pain Informed Movement and Pain Neuroscience Education | Standard Neuromuscular Exercise and OA Education
Number analyzed (Participants) | 28 | 31
score on a scale
  Baselin | 110.4 (23.7) | 102.2 (34.7)
  Follow-up | 120 (33.4) | 109.1 (32.2)

17. Other Pre Specified Outcome: Pain Intensity Measured on the Numeric Rating Scale (NRS)
Description: This outcome measure assesses pain intensity using the Numeric Rating Scale (NRS), where participants rate their pain on a scale from 0 to 10, with higher scores indicating greater pain severity. Three ratings are recorded: average pain intensity in the past 24 hours, average pain intensity in the past week, and worst pain intensity in the past 24 hours.
Time Frame: baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pain Informed Movement and Pain Neuroscience Education | Standard Neuromuscular Exercise and OA Education
Number analyzed (Participants) | 28 | 31
score on a scale
  Baseline Pain in the past 24 hours | 4.2 (1.7) | 3.5 (1.9)
  Baseline Pain in the past week | 4.2 (1.4) | 3.8 (1.9)
  Baseline worse pain in the past 24 hours | 4.9 (1.8) | 3.9 (2.4)
  Follow up Pain in the past 24 hours | 3.0 (2.2) | 2.8 (1.8)
  Follow-up Pain in the past week | 3.3 (1.6) | 3.1 (1.7)
  Follow up worse pain in the past 24 hours | 3.5 (2.7) | 3.2 (2.2)

18. Other Pre Specified Outcome: Pain Catastrophizing Scale (PCS)
Description: 13 questions for a total score of 52 with higher scores indicating more severe symptoms. Minimum score = 0, maximum score 52
Time Frame: baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pain Informed Movement and Pain Neuroscience Education | Standard Neuromuscular Exercise and OA Education
Number analyzed (Participants) | 28 | 31
score on a scale
  Baseline | 11.2 (9.6) | 9.4 (9.1)
  Follow-up | 7.4 (7.4) | 11.1 (6.8)

19. Other Pre Specified Outcome: Self-Efficacy for Managing Chronic Disease 6-item Scale (SEMCD-6)
Description: measure of self-efficacy rated on 0-10 scale ranging from not at all confident to entirely confident
Time Frame: baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pain Informed Movement and Pain Neuroscience Education | Standard Neuromuscular Exercise and OA Education
Number analyzed (Participants) | 28 | 31
score on a scale
  Baseline | 7.0 (1.5) | 6.8 (1.8)
  Follow-up | 7.4 (1.9) | 7.1 (2)

20. Other Pre Specified Outcome: Hospital Anxiety and Depression Scale (HADS)
Description: This outcome measure assesses symptoms of anxiety and depression using the Hospital Anxiety and Depression Scale (HADS). The HADS consists of 14 items, with seven items assessing anxiety (HADS-A) and seven assessing depression (HADS-D). Each item is scored on a 0 to 3 scale, resulting in total scores ranging from 0 to 21 for both anxiety and depression subscales.
  Higher scores indicate greater levels of anxiety or depression,
Time Frame: baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pain Informed Movement and Pain Neuroscience Education | Standard Neuromuscular Exercise and OA Education
Number analyzed (Participants) | 28 | 31
score on a scale
  Anxiety Baseline | 5.2 (3.2) | 4.9 (3.0)
  Depression Baseline | 3.6 (2.3) | 4.9 (3.0)
  Anxiety Follow-up | 5.2 (3.1) | 4.2 (3.6)
  Depression follow-up | 3.7 (2.3) | 3.8 (2.9)

21. Other Pre Specified Outcome: Brief Fear of Movement Scale for Osteoarthritis (BFMSO)
Description: This outcome measure assesses fear of movement (kinesiophobia) in individuals with osteoarthritis using the Brief Fear of Movement Scale for Osteoarthritis (BFMSO). The BFMSO consists of six items derived from the Tampa Scale for Kinesiophobia (TSK) and is rated on a 4-point Likert scale (1-4), with a total score range of 6 to 24, where higher scores indicate greater levels of kinesiophobia.
  The scale evaluates concerns about movement due to pain or the fear of worsening symptoms, providing insight into the psychological barriers that may affect physical activity and rehabilitation adherence in individuals with osteoarthritis.
Time Frame: Baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: Total score on a scale
Arm/Group | Pain Informed Movement and Pain Neuroscience Education | Standard Neuromuscular Exercise and OA Education
Number analyzed (Participants) | 28 | 31
Total score on a scale
  Baseline | 10.3 (2.7) | 10.4 (3.1)
  Follow-up | 11.8 (2.1) | 10.7 (3.1)

22. Other Pre Specified Outcome: Knee Injury and Osteoarthritis Outcome Score (KOOS)
Description: The KOOS pain and function in daily living and QoL subscales were used to assess self-reported opinions about patients' knee and associated problems. Scores ranged from 0-100 with zero representing extreme knee problems and 100 representing no knee problems
Time Frame: baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pain Informed Movement and Pain Neuroscience Education | Standard Neuromuscular Exercise and OA Education
Number analyzed (Participants) | 28 | 31
score on a scale
  Pain baseline | 55.3 (12.7) | 60.9 (14)
  Function baseline | 70.5 (12.1) | 71.2 (13.2)
  QL baseline | 23.6 (15.9) | 19.7 (16.8)
  Pain follow-up | 67.4 (13.5) | 57.7 (14.6)
  Function follow-up | 77.2 (12.1) | 76.7 (14.9)
  Ql- follow up | 28.1 (14) | 26.6 (15.2)

23. Other Pre Specified Outcome: Intermittent and Constant Osteoarthritis Pain (ICOAP) Knee Version
Description: The ICOAP (Intermittent and Constant Osteoarthritis Pain) Knee Version assesses two distinct types of knee pain: constant pain and intermittent pain. The constant pain subscale consists of five items that evaluate pain that is present all the time. Each item is rated on a scale from 0 to 4, where 0 represents no pain, 1 indicates mild pain, 2 corresponds to moderate pain, 3 signifies severe pain, and 4 represents extreme pain. The total score for this subscale ranges from 0 to 20, with higher scores reflecting greater pain severity.
  Similarly, the intermittent pain subscale comprises six items that assess pain that comes and goes in episodes. Each item follows the same 0 to 4 rating scale, capturing the intensity of episodic pain experiences. The total score for this subscale ranges from 0 to 24. The overall ICOAP knee score is the sum of both subscales, resulting in a total score range of 0 to 44, where higher scores indicate more severe and impactful knee pain.
Time Frame: baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Pain Informed Movement and Pain Neuroscience Education | Standard Neuromuscular Exercise and OA Education
Number analyzed (Participants) | 28 | 31
score on a scale
  Constant Pain - Baseline | 6.9 (3.3) | 5.5 (3.9)
  Intermittent Pain- Baseline | 10.2 (4.0) | 10.4 (3.6)
  Constant Pain - Follow-up | 4.4 (3.4) | 4.2 (3.7)
  Intermittent Pain- Follow up | 7.5 (4.2) | 7 (3.8)
  Total Score Baseline | 17.2 (6.3) | 16.1 (7.1)
  Total Score Follow up | 11.8 (7.3) | 11.1 (6.7)

24. Other Pre Specified Outcome: 30 Second Sit to Stand Test
Description: to measure functional leg strength and endurance by counting the numbers of complete movements accomplished in the allotted time
Time Frame: baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: repetitions
Arm/Group | Pain Informed Movement and Pain Neuroscience Education | Standard Neuromuscular Exercise and OA Education
Number analyzed (Participants) | 28 | 31
repetitions
  Baseline | 13.8 (3.3) | 11.9 (2.6)
  Follow-up | 17 (4) | 15 (4)

25. Other Pre Specified Outcome: Serum Levels of Brain Derived Neurotrophic Factors (BDNF) Via Blood Analysis
Description: a neurotrophin level measured in pg/ml
Time Frame: baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: picograms per milliliter
Arm/Group | Pain Informed Movement and Pain Neuroscience Education | Standard Neuromuscular Exercise and OA Education
Number analyzed (Participants) | 28 | 31
picograms per milliliter
  Baseline | 39.7 (8.9) | 39.3 (11.2)
  Follow-up | 40.3 (9) | 39.1 (10.2)

26. Other Pre Specified Outcome: Serum Levels of Nerve Growth Factor (NGF) Via Blood Analysis
Description: a neurotrophin level measured in pg/ml
Time Frame: baseline and 8 weeks
Measure: Mean (Standard Deviation); unit: picograms per milliliter
Arm/Group | Pain Informed Movement and Pain Neuroscience Education | Standard Neuromuscular Exercise and OA Education
Number analyzed (Participants) | 28 | 31
picograms per milliliter
  Baseline | 614 (1436) | 534 (1426)
  Follow-up | 587 (1460) | 521 (1564)

27. Other Pre Specified Outcome: Perspectives on the Effectiveness of the Different Intervention Components on Managing Pain
Description: One question will be asked of participants in each arm to rank the effectiveness of the different components of the intervention they received. e.g. "Please rank the different components of the intervention you received in order of how effective they are for managing your pain." A list of the different components in each study arm will be provided e.g. education videos, strengthening exercise, mind-body techniques
Time Frame: 8 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 8 weeks of the program
Description: The study design not including long-term mortality tracking.
Arm/Group | Pain Informed Movement and Pain Neuroscience Education | Standard Neuromuscular Exercise and OA Education
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/35
Other Adverse Events (participants affected / at risk) | 0/34 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-03): https://cdn.clinicaltrials.gov/large-docs/29/NCT05730829/Prot_SAP_000.pdf
  • Informed Consent Form (2023-02-06): https://cdn.clinicaltrials.gov/large-docs/29/NCT05730829/ICF_001.pdf